CLINICAL TRIAL: NCT06407882
Title: Effects pf Conductive Exercises on Motor Skills Among the Children With Cerebral Palsy
Brief Title: Effects of Conductive Exercises on Motor Skills Among the Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07103
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: ADLS,; Cerebral palsy,; Motor skills,; Quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be Randomized control trial in which non probabilty convenient sampling will be used. Two groups of 6-12 age will be formed in which participants will be randomly divided. Group A will only receive Conductive education and group B will receive conventional physical therapy.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Group A will perform Conductive exercises (CE) in addition to routine physical therapy. Conductive exercises program will include Squat-position, Rising from squat to stand, Sitting on the stool, Prone lying, High kneeling and half kneeling, Sitting, lying and high kneeling, Walking in parallel bars, Sitting to standing, Floor to standing, Picking up toys from the floor, Balance on one foot on different surfaces and heights, Crawling over foams of different sizes and shapes, Climbing steps or stairs sometimes while carrying a toy. These exercises will improve motor skills and activities of daily living by improving the muscle strength
  Interventions: Behavioral: Conductive Exercises
- Routine Physical Therapy (Active Comparator): Group B will perform routine physical therapy (RPT) alone. Active and passive movements, Passive stretching, strengthening exercises, weight bearing exercises.
  Interventions: Behavioral: Routine Physical Therapy

INTERVENTIONS:
Behavioral: Conductive Exercises — Conductive education (CE) is a useful educational system for the management of motor disabled individuals whose disability and dysfunction was due to the damage to the central nervous system, mainly at the pre-, peri- or post-natal period of life. Conductive exercises basically include task-oriented learning within highly structured programs and conductors who are trained in special education and therapy administer the conductive education program
  Arms: Experimental Group
Behavioral: Routine Physical Therapy — Group B will perform routine physical therapy (RPT) alone. Active and passive movements, Passive stretching, strengthening exercises, weight bearing exercises.
  Arms: Routine Physical Therapy

SUMMARY:
Cerebral palsy (CP) is defined as a neurodevelopmental disorder in which there are abnormalities of motor skills, muscle tone ,and, movement and is caused by injury to the developing brain. Risk factors for cerebral palsy are most probably intrauterine exposure to infection or inflammation and disorders of coagulation.Cerebral palsy (CP) is classified as Spastic, Athetoid, Tremor, Rigidity, Ataxic, Atonic, and Mixed.

Cerebral Palsy (CP) is the most common cause of physical disability in early childhood and overall, the CP rate is between 2 and 3 per 1000 live births.There are several interventions to manage cerebral palsy depending upon the severity and type of cerebral palsy and hence requires a multidisciplinary setting for proper improvement and management.One of the important intervention is conductive education including conductive exercises (CE).

Conductive education (CE) is a useful educational system for the management of motor disabled individuals whose disability and dysfunction was due to the damage to the central nervous system, mainly at the pre-, peri- or post-natal period of life. Conductive exercises basically include task-oriented learning within highly structured programs and conductors who are trained in special education and therapy administer the conductive education program.

DETAILED DESCRIPTION:
Group A: Experimental group:

Group A will perform Conductive exercises (CE) in addition to routine physical therapy. Conductive exercises program will include Squat-position, Rising from squat to stand, Sitting on the stool, Prone lying, High kneeling and half kneeling, Sitting, lying and high kneeling, Walking in parallel bars, Sitting to standing, Floor to standing, Picking up toys from the floor, Balance on one foot on different surfaces and heights, Crawling over foams of different sizes and shapes, Climbing steps or stairs sometimes while carrying a toy. These exercises will improve motor skills and activities of daily living by improving the muscle strength.

Group B: Control group:

Group B will perform routine physical therapy (RPT) alone. Active and passive movements, Passive stretching, strengthening exercises, weight bearing exercises.

Both the groups will receive intervention for 45 minutes per session 5 days in a week for 2 month. Data will be collected at baseline and after the completion of the study. Data will be collected after ethical approval and consent. All the personal information of the patient will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Spastic cerebral palsy
* GMFCS level I, II and III
* Age group 6 to 12 years
* Either gender

Exclusion Criteria:

* Had a botulinum injection for reduce spasticity
* Subjects with any cardiac problem(congenitally)
* Children who are having visual and hearing deficits

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Gross motor function measure-88 (GMFM-88) | 8 weeks
  The Gross Motor Function Measure-88 (GMFM88) is a tool which is used to measure changes in gross motor function in cerebral palsy children and has been commonly used by researchers .The GMFM-88 consists of 88 items in five dimensions which are lying and rolling (GMFM-A); sitting (GMFM-B); crawling and kneeling (GMFM-C); standing (GMFM-D); and walking, running and jumping (GMFM-E).The psychometric properties of the adapted GMFM-88 for children with CP are reliable.
Cerebral Palsy Quality of Life Questionnaire (CP QOL) | 8 weeks
  The Cerebral Palsy Quality of Life for Children (CP QOL-Child) was made to assess several aspects of subjective happiness and well-being, rather than ill-being or functioning. It is productive to establish a profile of qualify of life of cerebral palsy children to understand their subjective perception of their life.The reliability and validity of the CP QOL-Child have been established, including internal consistency, test-retest reliability, and construct validity
ABILHAND questionnaire | 8 weeks
  This questionnaire is used to evaluate the effects of interventions that are useful for improving functional limitations under the different contextual situations.This is a valid and reliable assessment method which is used to assess a child's both unimanual and bimanual upper limb activities.This questionnaire focuses on the child's manual performance of 21 daily activities as perceived by the parents

CONTACTS AND LOCATIONS:
Overall Officials: Moneeza Ahmad, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulati S, Sondhi V. Cerebral Palsy: An Overview. Indian J Pediatr. 2018 Nov;85(11):1006-1016. doi: 10.1007/s12098-017-2475-1. Epub 2017 Nov 20. PMID 29152685